CLINICAL TRIAL: NCT00326248
Title: A Phase III, Multicenter, Randomized, Double-blind, Parallel Group Study to Evaluate the Safety and Efficacy of 50mg Oral Dosing With the Neurokinin-1 Receptor Antagonist GW679769 for the Prevention of Postoperative Nausea and Vomiting in Female Subjects at High Risk for Emesis
Brief Title: Casopitant (Oral) And ZOFRAN To Prevent Postoperative Nausea And Vomiting In Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NKT102553
Record Dates: First submitted 2006-05-12; First posted 2006-05-16 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Nausea and Vomiting, Postoperative
Keywords: postoperative nausea and vomiting PONV antiemetics NK-1 5HT3 casopitant mesylate ZOFRAN ondansetron hydrochloride
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — casopitant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: GW679769 (casopitant)

INTERVENTIONS:
Drug: GW679769 (casopitant)

SUMMARY:
This study is being conducted to see if adding GW679769 (casopitant) to ZOFRAN will significantly decrease the number of patients who experience nausea and vomiting after surgery.

ELIGIBILITY:
Inclusion criteria:

* History of PONV and/or motion sickness.
* Have not smoked for the last 6 months.
* Having certain types of abdominal, breast or shoulder surgeries.

Exclusion criteria:

* Pregnant or breastfeeding.
* Taking certain medications.
* Have certain pre-existing medical conditions.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 482 (Actual)
Dates: Start 2006-03; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Rates of vomiting and retching | after surgery

SECONDARY OUTCOMES:
Rates of nausea. Blood test results. | after surgery

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (53):
- United States (23):
  - GSK Investigational Site, Montgomery, Alabama
  - GSK Investigational Site, Sheffield, Alabama
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Boynton Beach, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Melbourne, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Naples, Florida
  - GSK Investigational Site, Pensacola, Florida
  - GSK Investigational Site, Anderson, Indiana
  - GSK Investigational Site, Grand Rapids, Michigan
  - GSK Investigational Site, Jackson, Mississippi
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, New Brunswick, New Jersey
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Altoona, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Spokane, Washington
- Canada (5):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Charlottetown, Prince Edward Island
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Regina, Saskatchewan
- France (7):
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Caen
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Rennes
  - GSK Investigational Site, Riom
  - GSK Investigational Site, Strasbourg
- Germany (3):
  - GSK Investigational Site, Marburg, Hesse
  - GSK Investigational Site, Aachen, North Rhine-Westphalia
  - GSK Investigational Site, Koblenz, Rhineland-Palatinate
- Hong Kong (2):
  - GSK Investigational Site, Pokfulam
  - GSK Investigational Site, Shatin, New Territories
- Hungary (4):
  - GSK Investigational Site, Győr
  - GSK Investigational Site, Miskolc
  - GSK Investigational Site, Szentes
  - GSK Investigational Site, Székesfehérvár
- Ireland (2):
  - GSK Investigational Site, Dublin
  - GSK Investigational Site, Galway
- GSK Investigational Site, Karachi, Pakistan
- Philippines (2):
  - GSK Investigational Site, Manila
  - GSK Investigational Site, Santa Cruz, Manila
- GSK Investigational Site, Bangkok, Thailand
- United Kingdom (3):
  - GSK Investigational Site, Glasgow, Lanarkshire
  - GSK Investigational Site, Livingston, West Lothian
  - GSK Investigational Site, Liverpool

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Altorjay A, Melson T, Chinachoit T, Kett A, Aqua K, Levin J, Blackburn LM, Lane S, Pergolizzi JV Jr. Casopitant and ondansetron for postoperative nausea and vomiting prevention in women at high risk for emesis: a phase 3 study. Arch Surg. 2011 Feb;146(2):201-6. doi: 10.1001/archsurg.2010.327. PMID 21339433
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: NKT102553 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: NKT102553 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: NKT102553 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: NKT102553 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: NKT102553 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: NKT102553 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: NKT102553 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register